CLINICAL TRIAL: NCT03946046
Title: Results of Botulinum Toxin Injections for Cervical Dystonia : Benefits of Ultrasonography
Brief Title: Targeting Methods of Botulinum Toxin Injections for Cervical Dystonia
Acronym: RINOCERAUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2017_68; 2018-A02045-50 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2019-04-26; First posted 2019-05-10 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Idiopathic Cervical Dystonia
Keywords: Cervical dystonia; Botulinum toxin; Ultrasound-guided injection; CDIP58; TWSTRS-2
MeSH Terms: conditions — Torticollis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical targeting (Experimental): Clinical localization method (observation and palpation of target muscles)
  Interventions: Procedure: Clinical targeting
- Ultrasonography targeting (Experimental): Ultrason-guided method
  Interventions: Procedure: Ultrasonography targeting

INTERVENTIONS:
Procedure: Clinical targeting — The intervention consists of the injection of botulinum toxin A into muscles targeted by a clinical localization method (observation and palpation of target muscles)
  Arms: Clinical targeting
Procedure: Ultrasonography targeting — The intervention consists of the injection of botulinum toxin A into muscles by ultrason-guided method
  Arms: Ultrasonography targeting

SUMMARY:
Botulinum toxin injections are the treatment of choice for cervical dystonia. Even if this treatment is successful for most of the patients, partials or completes failures still remained.

Usually, botulinum toxin injections are realized by clinical localization techniques (observation and palpation of target muscles). The use of Ultrasonography to guide injections of Botulinum toxin has theoretical benefits (as an improved precision, an improved reproducibility, the targeting of deep-seated muscles, and a lower risk of adverse events) but its interest has never been demonstrated.

DETAILED DESCRIPTION:
Open label non-randomised controlled clinical trial comparing clinical localization techniques and ultrasonography to guide injections of Botulinum toxin A.

The primary outcome is to compare both techniques of injection regarding to the health impact of cervical dystonia (CDIP-58) measured 1 month after injection.

The results of this clinical trial will help the clinician to decide which strategy of injection is the most effective in terms of benefit/risk ratio to treat the cervical dystonia.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18 years old
* Focal idiopathic cervical dystonia treated by injections of Botulinum toxin type A (onabotulinumtoxinA, Botox® ; abobotulinumtoxinA, Dysport® ; or incobotulinumtoxinA, Xeomin®).
* Patient who have previously received at least 3 cycles of botulinum toxin A injections in this specific indication
* Injections realized with clinical targeting exclusively or ultrasonography targeting exclusively
* Patient who is not opposed to its participation in this study
* Patient affiliated to the Sécurité Sociale
* Patient able to comply with study procedures and study duration

Exclusion Criteria:

* Woman pregnant, woman of childbearing age not taking effective contraception or breastfeeding
* Contraindication of botulinum toxin injections as :

  * Hypersensivity to the botulinum toxin A or to an excipient of the commercialized treatment (onabotulinumtoxinA, Botox® ; abobotulinumtoxinA, Dysport® ; incobotulinumtoxinA, Xeomin®)
  * Generalized muscular activity disorder (Myasthenia gravis, Lambert-Eaton syndrome)
  * Infection or inflammation of the injection site
* Concomitant treatment that can interact with botulinum toxin A or modify the function of the neuromuscular synapse junction (anticholinergics, curare and other myorelaxing agents, Aminoglycosides, amino-4-quinolines)
* Documented resistance to the botulinum toxin A
* Inability to receive the information, inability to participate to the all study duration, refusal to sign the consent
* EMG-guided botulinum toxin injections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2020-04-14 (Actual); Study Completion 2020-04-14 (Actual)

PRIMARY OUTCOMES:
Cervical Dystonia Impact Profile 58 (CDIP-58) | 1 month after inclusion
  Variation of the total score obtained with The Cervical Dystonia Impact Profile

SECONDARY OUTCOMES:
Placement of the injecting needle | the day of the inclusion
  Assessment of the accurate placement of the injecting needle within the target muscle by ultrasonography in patients injected by the clinical targeting method (number and percent of discordances)
GCI-I (Clinical Global Impressions - Improvement) patient scale | 1 month after inclusion
  Variation of the GCI-I (Clinical Global Impressions - Improvement) patient scale :
  1. = Very much improved : nearly all better; good level of functioning; minimal symptoms; represents a very substantial change
  2. = Much improved : notably better with significant reduction of symptoms; increase in the level of functioning but some symptoms remain
  3. = Minimally improved : slightly better with little or no clinically meaningful reduction of symptoms. Represents very little change in basic clinical status, level of care, or functional capacity
  4. = No change : symptoms remain essentially unchanged
  5. = Minimally worse : slightly worse but may not be clinically meaningful; may represent very little change in basic clinical status or functional capacity
  6. = Much worse : clinically significant increase in symptoms and diminished functioning
  7. = Very much worse : severe exacerbation of symptoms and loss of functioning
TWSTRS-2 (Toronto Western Spasmodic Torticollis Rating Scale) : pain scale only | 1 month after inclusion
  Variation of the TWSTRS-2 (Toronto Western Spasmodic Torticollis Rating Scale) : pain scale only
  Total score = 0 (no pain) to 40 (maximal pain)
TWSTRS-PSYCH (Toronto Western Spasmodic Torticollis Rating Scale - Psychiatric) scale | 1 month after inclusion
  Variation of the TWSTRS-PSYCH (Toronto Western Spasmodic Torticollis Rating Scale - Psychiatric) scale
  Total score = 0 (no psychiatric disorders) to 24 (important psychiatric disorders)
Rate of Adverse Events | 1 month after inclusion
  Adverse events related to the botulinum toxin injection (pain, swallowing disorders, hematoma, muscular weakness, dry mouth)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre KREISLER, MD, Ph, Principal Investigator — Hôpital Roger Salengro, CHRU Lille
Locations (1):
- Hôpital Roger Salengro, CHRU de Lille - Service de neurologie A, Lille, France